CLINICAL TRIAL: NCT03396367
Title: Intervention to Reduce Drug Use and HIV Incidence Among High PrEP Priority Partnered YMSM
Brief Title: Prevention and Risk: Treatment With a New Emphasis on Relationships
Acronym: PARTNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tyrel Starks, Professor of Psychology, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA045613 (NIH); R01DA045613 (NIH)
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Adherence, Medication; Risk Reduction; Drug Use; Sex, Anal; HIV/AIDS
Keywords: Relationships; YMSM; HIV/AIDS; PrEP; Drug Use
MeSH Terms: conditions — Medication Adherence; Risk Reduction Behavior; Sexual Behavior; Acquired Immunodeficiency Syndrome | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARTNER Intervention (Experimental): This intervention is a four-session intervention designed to increase PrEP uptake, increase PrEP adherence, and reduce drug use and HIV transmission risk behaviors of individuals in relationships.
  Interventions: Behavioral: PARTNER
- Education Intervention (Active Comparator): This intervention is a four-session intervention that discussed drug use and its effect on physiological social functioning.
  Interventions: Behavioral: Education Intervention

INTERVENTIONS:
Behavioral: PARTNER — The PATRNER intervention addresses, drug use, PrEP uptake/adherence, and HIV transmission risk by enhancing communication skills by integrating motivational interviewing and video-based communication skills training.
  Arms: PARTNER Intervention
Behavioral: Education Intervention — The Education intervention consists of a 4-session health education intervention that addresses sexual risk and substance use through a lecture and question and answer format.
  Arms: Education Intervention

SUMMARY:
This research examines the efficacy of an individually-delivered intervention tailored for YMSM in relationships. The intervention - termed PARTNER - utilizes a brief (4 session) motivational interviewing format to target Pre-Exposure Prophylaxis (PrEP) uptake/adherence, HIV transmission risk behavior, and associated drug use.

DETAILED DESCRIPTION:
This study aims to evaluate a individual-focused intervention with an integrated focus on drug use and HIV prevention, including uptake of and adherence to PrEP. The investigators will recruit a sample of 240 partnered individuals.

Recruitment occurs using a mix of in-person and Internet recruitment. Outreach workers will visit bars and events in the New York City area to recruit participants. Also,information on our project will be posted on social media sites (e.g.,Facebook, Grindr, Scruff). Interested individuals will complete a brief online screener to assess eligibility. A telephone screener will be conducted with participants who are preliminarily eligible based upon online screener responses. Participants who are eligible based upon telephone screening responses will be sent an email. The email contains a link for them to access the baseline online survey. It provides information which introduces the study to the recruited partner and a link to the baseline survey online. If participants indicate intimate partner violence (IPV) on the online baseline survey, participants will be rendered ineligible. Only the participant that indicated experiencing IPV will be given a list of local referrals to access IPV-related services.

An in-person baseline assessment appointment will be scheduled after both participants have completed the online survey.

The in-person baseline assessment appointment consists of four components; written consent, a computer-assisted self interview (CASI), a timeline follow back interview, and biological testing.

Written consent is obtained prior to the start of any in-person baseline activity. Participants additionally complete a computer-assisted self interview (CASI). After this, participants will independently complete a TFLB. TLFB is a semi-structured interview to collect retrospective event-level data on drug use, sexual behavior and PrEP adherence (for those on PrEP) in the past 30 days.

The final part of the in-person baseline assessment consists of biological testing for STI (gonorrhea & chlamydia via urinalysis and rectal swabs), drug testing via 5-panel fingernail drug assay via finger or toe nail clippings. Drugs tested are 5 major drugs: Amphetamines, Cannabinoids, Cocaine, Opiates, and Phencyclidine (PCP). HIV testing will consist of a finder prick test using the Alere Determine HIV-1/2 Ag/Ab Combo test. Participants indicating current PrEP use will receive an HIV test via blood draw for a laboratory immunoassay. Participants indicating current PrEP give an additional blood sample and fingernail sample to examine PrEP adherence using a dried blood spot for western blot analysis and fingernail assay.

After the baseline assessment, participants will be randomized to receive their first PARTNER or Education session, of which will occur immediately following their baseline assessment.

The study will employ a stratified randomization procedure using an algorithm via Qualtrics. Participants will be randomized using three couple-level criteria as reported by the participant. Participants will be randomized based on relationship length difference (less than 2 years versus 2 or more), age difference (less than 3 years versus 3 or more), racial difference (both white versus all others combinations), PrEP use (Participant reports current PrEP use versus does not report current use).

Each of the intervention arms consists of 4 sessions that occur once a week for four consecutive weeks.

All participants complete a 3-month, 6-month, 9-month, and 12-month follow ups. At the 3 month follow up (post baseline assessment), participants complete a survey with a TLFB, fingernail specimen collection for drug use. For participants indicating current PrEP use, participants and give blood for a dried blood spot analysis and an additional fingernail sample to test for PrEP uptake/adherence.

At the 6 month follow up month follow up (post baseline assessment), participants complete a survey with a TLFB, fingernail specimen collection for drug use, biological testing for STI (gonorrhea & chlamydia via urinalysis and rectal swabs) and HIV testing using the Alere Determine HIV-1/2 Ag/Ab Combo test. Participants indicating current PrEP use will receive an HIV test via blood draw for a laboratory immunoassay Also, for participants indicating current PrEP use, participants and give blood for a dried blood spot analysis and an additional fingernail sample to test for PrEP uptake/adherence.

At the 9 month follow up (post baseline assessment), participants complete a survey with a TLFB, fingernail specimen collection for drug use. For participants indicating current PrEP use, participants and give blood for a dried blood spot analysis and an additional fingernail sample to test for PrEP uptake/adherence.

At final assessment (12 month follow up post baseline assessment), participants complete a survey with a TLFB, fingernail specimen collection for drug use, biological testing for STI (gonorrhea & chlamydia via urinalysis and rectal swabs) and HIV testing using the Alere Determine HIV-1/2 Ag/Ab Combo test. Participants indicating current PrEP use will receive an HIV test via blood draw for a laboratory immunoassay Also, for participants indicating current PrEP use, participants and give blood for a dried blood spot analysis and an additional fingernail sample to test for PrEP uptake/adherence.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 29 years of age (inclusive);
* Main partner must be aged 18 or older.
* Must be in a main partner relationship with another male (duration ≥ 1 months);
* HIV-negative serostatus (confirmed by rapid test);
* Recent (past 30 day) use of at least one of the substances identified as most commonly used by YMSM (marijuana, cocaine, methamphetamine, heroin or other opiates, MDMA, psychedelics, GHB, and/or ketamine);
* Sexual behavior meeting CDC criteria for PrEP candidacy (TRB with a casual partner in the past 30 days or TRB with a non-monogamous or serodiscordant main partner).
* Participants must reside in the NYC metro area
* Ability to communicate in English

Exclusion Criteria:

* Unstable, serious psychiatric symptoms (assessed by the Psychotic Disorder subsection of the Structured Clinical Interview for DSM-IV);
* Current suicidal/homicidal ideation;
* Evidence of gross cognitive impairment (a score of <24 on the mini-mental state examination)
* A history of severe physical or sexual Intimate Partner Violence (IPV) victimization in the current relationship in which participants report not currently feeling "safe" in their relationship and/or coerced to participate in the study.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both gender at birth and current self-identified gender must be male.
Enrollment: 196 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyrel J Starks, PhD, Principal Investigator — Hunter College of City University of New York
Locations (1):
- Hunter College- City University of New York, New York, New York, United States

REFERENCES:
- [Background] Parsons JT, Lelutiu-Weinberger C, Botsko M, Golub SA. A randomized controlled trial utilizing motivational interviewing to reduce HIV risk and drug use in young gay and bisexual men. J Consult Clin Psychol. 2014 Feb;82(1):9-18. doi: 10.1037/a0035311. Epub 2013 Dec 23. PMID 24364800
- [Derived] Starks TJ, Robles G, Pawson M, Jimenez RH, Gandhi M, Parsons JT, Millar BM. Motivational Interviewing to Reduce Drug Use and HIV Incidence Among Young Men Who Have Sex With Men in Relationships and Are High Priority for Pre-Exposure Prophylaxis (Project PARTNER): Randomized Controlled Trial Protocol. JMIR Res Protoc. 2019 Jul 4;8(7):e13015. doi: 10.2196/13015. PMID 31274114

RESULTS

PARTICIPANT FLOW:
Groups:
- Partner Intervention: The PATRNER intervention addresses, drug use, PrEP uptake/adherence, and HIV transmission risk by enhancing communication skills by integrating motivational interviewing and video-based communication skills training.
Period: Overall Study
Arm/Group | Partner Intervention | Education Intervention
Started | 94 | 102
Completed | 94 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Partner Intervention | Education Intervention | Total
Number analyzed (Participants) | 94 | 102 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (2.8) | 27 (2.8) | 26.9 (2.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender Male | 94 | 102 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 53 | 47 | 100
  Black or African American | 6 | 5 | 11
  Latino or Hispanic | 23 | 31 | 54
  Asian, Pacific Islander | 6 | 10 | 16
  Multiracial or another identity | 6 | 9 | 15
Sexual Identity [Count of Participants; unit: Participants]
  Gay | 70 | 88 | 158
  Bisexual | 10 | 8 | 18
  Queer or another Identity | 13 | 5 | 18
  unknown | 1 | 1 | 2
Region of Residence [Count of Participants; unit: Participants]
  Northeast | 83 | 95 | 178
  Elsewhere in the US | 11 | 7 | 18
Education [Count of Participants; unit: Participants]
  Less than a 4 year degree | 19 | 24 | 43
  4 year degree or higher | 74 | 77 | 151
  unknown | 1 | 1 | 2
PrEP status [Count of Participants; unit: Participants]
  Not taking PrEP | 44 | 44 | 88
  Current PrEP perscription | 50 | 58 | 108
Interpersonal Communication Communication Competence Scale [Mean (Standard Deviation); unit: units on a scale] — The Interpersonal Communication Competence Scale (Rubin, 1994) assesses self-disclosure, social anxiety, assertiveness, and empathy. Each statement is evaluated on a 5- point Likert scale ranging from 0 (almost never) to 4 (almost always). Total score was summed and had a range of 0 to 48. Higher scores indicated greater communication competence.
  Rubin RB, Martin MM. Development of a measure of interpersonal competence. Communication Research Reports. 1994;11(1):33-44.
  units on a scale | 43.3 (5.9) | 44.4 (5.9) | 43.8 (5.9)
Approximation to an Ideal subscale of the Multiple Determinants of Relationship Commitment Inventory [Mean (Standard Deviation); unit: units on a scale] — Relationship satisfaction is assessed using the approximation to ideal subscale of the Multiple Determinants of Relationship Commitment Inventory (Kurdek, 1998). The subscale is 4 items with response options ranging from 1 (strongly disagree) to 5 (strongly agree). Total range is 4 to 20. Higher scores indicated greater relationship satisfaction.
  Kurdek LA. Relationship outcomes and their predictors: Longitudinal evidence from heterosexual married, gay cohabiting, and lesbian cohabiting couples. Journal of Marriage and the Family. 1998;60(3):553-68.
  units on a scale | 15.1 (3.7) | 15.4 (3.1) | 15.2 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Illicit Drug Use Days
Description: The self-reported number of illicit drug use days (not including marijuana) in the past 30 days
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Partner Intervention | Education Intervention
Number analyzed (Participants) | 94 | 102
days
  Baseline | 1.49 (5.37) | .80 (2.14)
  3-month | 1.16 (3.83) | 0.83 (2.3)
  6-month | .67 (1.79) | .56 (1.29)
  9-month | 1.08 (3.62) | .81 (2.30)
  12-month | .66 (1.49) | .67 (1.55)
Statistical Analysis 1: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .433, Latent Growth Curve — Condition (referent = education control); Slope = .372, 95% CI 2-sided [-.558 to 1.302] — Variable:
Statistical Analysis 2: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .749, Latent Growth Curve; Slope = -.017, 95% CI 2-sided [-.121 to .087] — Variable: Communication Compentence
Statistical Analysis 3: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .302, Latent Growth Curve; Slope = .073, 95% CI 2-sided [-.121 to .087] — Moderating Variable: Communication Competence by Condition
Statistical Analysis 4: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .799, Latent Growth Curve; Slope = .027, 95% CI 2-sided [-.182 to .236] — Variable: Relationship Satisfaction
Statistical Analysis 5: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .173, Latent Growth Curve; Slope = -.211, 95% CI 2-sided [-.514 to .092] — Moderating Variable: Relationship Satisfaction by Condition

2. Primary Outcome: Cannabis Use Days
Description: The self-reported number of cannabis drug use days in the past 30 days
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Partner Intervention | Education Intervention
Number analyzed (Participants) | 94 | 102
days
  Baseline | 9.68 (11.25) | 7.59 (10.64)
  3-Month | 9.28 (11.58) | 7.49 (10.33)
  6-Month | 9.13 (11.63) | 7.27 (10.39)
  9-Month | 10.04 (12.24) | 6.88 (10.73)
  12-Month | 10.04 (12.55) | 6.61 (10.64)
Statistical Analysis 1: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .172, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between the Partner intervention and the Education intervention at baseline; Slope = .427, 95% CI 2-sided [-.186 to 1.04]
Statistical Analysis 2: Comparison: Partner Intervention; Test type: Superiority; p = .054, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between the Partner intervention and the Education intervention at the 3-month follow-up; Slope = -.281, 95% CI 2-sided [-.623 to .061]
Statistical Analysis 3: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .036, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between the Partner intervention and the Education intervention across the 3-,6-,9-, and 12- month follow-ups; Slope = 0.125, 95% CI 2-sided [-.011 to .260]

3. Primary Outcome: Number (Proportion) of Participants Who Report Sexual HIV Transmission Risk With Casual Partners
Description: The percentage of participants in each condition reporting sexual HIV transmission risk with a casual partner (any condomless sex with a casual partner in the absence of PrEP).
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month
Population: intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Partner Intervention | Education Intervention
Number analyzed (Participants) | 94 | 102
Participants
  Baseline | 16 | 16
  3-Month | 8 | 10
  6-Month | 5 | 5
  9-Month | 6 | 6
  12-Month | 11 | 12
Statistical Analysis 1: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .679, Latent Growth Curve — [p-value comment as in outcome 2, analysis 1]; Slope = .245, 95% CI 2-sided [-.913 to 1.403]
Statistical Analysis 2: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .359, Latent Growth Curve — [p-value comment as in outcome 2, analysis 2]; Slope = -.301, 95% CI 2-sided [-1.938 to 1.336]
Statistical Analysis 3: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .431, Latent Growth Curve — [p-value comment as in outcome 2, analysis 3]; Slope = .048, 95% CI 2-sided [-.496 to .593]

4. Primary Outcome: The Number (Proportion) of Participants Reporting Pre-Exposure Prophylaxis (PrEP) Uptake
Description: The percentage participants in each condition who report having a current PrEP prescription at the time of follow-up.
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month,
Population: intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Partner Intervention | Education Intervention
Number analyzed (Participants) | 94 | 102
Participants
  Baseline | 50 | 58
  3-Month | 42 | 51
  6-Month | 50 | 47
  9-Month | 52 | 45
  12-Month | 43 | 46
Statistical Analysis 1: Comparison: Partner Intervention; Test type: Superiority; p = .326, Latent Growth Curve — [p-value comment as in outcome 2, analysis 1]; Slope = -1.251, 95% CI 2-sided [-3.814 to 1.311]
Statistical Analysis 2: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .384, Latent Growth Curve — [p-value comment as in outcome 2, analysis 2]; Slope = .246, 95% CI 2-sided [-1.383 to 1.875]
Statistical Analysis 3: Comparison: Partner Intervention vs Education Intervention; Test type: Superiority; p = .019, Latent Growth Curve — [p-value comment as in outcome 2, analysis 3]; Slope = .856, 95% CI 2-sided [.052 to 1.659]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | PARTNER Intervention | Education Intervention
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/102
Other Adverse Events (participants affected / at risk) | 0/94 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03396367/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03396367/ICF_001.pdf